CLINICAL TRIAL: NCT03865212
Title: Phase I Trial to Evaluate the Safety and Efficacy of Intratumoral and Intravenous Injection of Vesicular Stomatitis Virus Expressing Human Interferon Beta and Tyrosinase Related Protein 1 (VSV-IFNb-TYRP1) in Patients With Metastatic Ocular Melanoma and Previously Treated Patients With Unresectable Stage III/IV Cutaneous Melanoma
Brief Title: Modified Virus VSV-IFNbetaTYRP1 in Treating Patients With Stage III-IV Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding; lack of objective response
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1376; NCI-2019-01127 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1376 (Other: Mayo Clinic in Florida); 18-000991 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Choroid Melanoma; Metastatic Melanoma; Metastatic Mucosal Melanoma; Metastatic Uveal Melanoma; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Unresectable Melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — TYRP1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (VSV-IFNbetaTYRP1) (Experimental): Patients receive recombinant vesicular stomatitis virus-expressing interferon-beta and tyrosinase related protein 1 IT and IV over 30-60 minutes 2-4 hours later on day 1.
  Interventions: Drug: Recombinant Vesicular Stomatitis Virus-expressing Interferon-beta and Tyrosinase Related Protein 1
- Group B (VSV-IFNbetaTYRP1) (Experimental): Patients receive recombinant vesicular stomatitis virus-expressing interferon-beta and tyrosinase related protein 1 IT and IV over 30-60 minutes 2-4 hours later on day 1. Cycle 1 continues for 28 days, with subsequent cycles repeating every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Recombinant Vesicular Stomatitis Virus-expressing Interferon-beta and Tyrosinase Related Protein 1

INTERVENTIONS:
Drug: Recombinant Vesicular Stomatitis Virus-expressing Interferon-beta and Tyrosinase Related Protein 1 — Given IT and IV
  Other Names: Recombinant VSV-expressing IFN-b and TYRP1; Recombinant VSV-IFNbetaTYRP1; VSV-IFN-b/TYRP1; VSV-IFNbetaTYRP1

SUMMARY:
This phase I trial studies the side effects and best dose of a modified virus called VSV-IFNbetaTYRP1 in treating patients with stage III-IV melanoma. The vesicular stomatitis virus (VSV) has been altered to include two extra genes: human interferon beta (hIFNbeta), which may protect normal healthy cells from becoming infected with the virus, and TYRP1, which is expressed mainly in melanocytes (specialized skin cell that produces the protective skin-darkening pigment melanin) and melanoma tumor cells, and may trigger a strong immune response to kill the melanoma tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety profile and maximum tolerated dose (MTD) of recombinant vesicular stomatitis virus-expressing interferon-beta and tyrosinase related protein 1 (VSV-IFNbeta-TYRP1) therapy when administered by intravenous (IV) and intratumoral (IT) injection in patients with previously treated metastatic melanoma.

SECONDARY OBJECTIVE:

I. To gather preliminary data on tumor response rate and progression-free survival time of VSV-IFNbeta-TYRP1 intravenous and intratumoral therapy among patients with metastatic malignant melanoma.

CORRELATIVE OBJECTIVES:

I. To determine the pharmacokinetic (PK) profile of VSV-IFNbeta-TYRP1 in patients by measurement of viremia in the blood using reverse transcriptase polymerase chain reaction (RT-PCR) for VSV-N ribonucleic acid (RNA).

II. To characterize the pharmacodynamics (PD) of VSV-IFNbeta-TYRP1 by measuring serum interferon-beta.

III. To determine if there is viral shedding (mouthwash, buccal swab, and urine) before and after viral treatment at different time points.

IV. Assess fresh pre- and post-treatment tumor biopsy samples for viral RNA, viral protein by immunohistochemistry (IHC), infectious virus recovery, infiltrating immune cells.

V. Assess transcriptome of fresh pre- and post-treatment tumor biopsy samples. VI. Assess exome of fresh peripheral blood lymphocytes (PBL) and fresh tumor samples pre-VSV treatment for neoantigen profiling.

VII. Assess changes in cytokine levels and immune cell profile in peripheral blood and tumor samples, pre and post viral treatment.

VIII. Assess if there is an increase in the amount of VSV and melanoma antigen, specifically TYRP1, reactive IFN-gamma secreting T cells by intracellular staining intracellular cytokine (ICS) and enzyme-linked immunosorbent spot (ELISpot) assays.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 groups.

GROUP A: Patients receive recombinant vesicular stomatitis virus-expressing interferon-beta and tyrosinase related protein 1 intratumorally (IT) and intravenously (IV) over 30-60 minutes 2-4 hours later on day 1.

GROUP B: Patients receive recombinant vesicular stomatitis virus-expressing interferon-beta and tyrosinase related protein 1 IT and IV over 30-60 minutes 2-4 hours later on day 1. Cycle 1 continues for 28 days, with subsequent cycles repeating every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients in Group A are followed up at 42 days. Patients in Group B are followed up at 28 days, every 3 months until progressive disease, and then every 6 months for a maximum of 5 years after study registration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histologically or cytologically confirmed diagnosis of unresectable stage III or metastatic (stage IV) melanoma, including metastatic ocular melanoma
* Cutaneous melanoma patients only:

  * At least one prior Food and Drug Administration (FDA) approved systemic therapy in the metastatic setting; and disease progression after immune checkpoint inhibitors
  * If tumor is BRAF-mutated, previous BRAF- and/or MEK-targeted therapies are required
  * NOTE: for ocular melanoma patients no current standard of care exists, so patients are permitted to be treated in 1st line setting
* Measurable disease by any imaging modality as defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1)

  * NOTE: disease that is measurable by physical examination only is not eligible
* Injectable disease (i.e., suitable for direct injection or through the use of ultrasound guidance) defined as:

  * At least 1 injectable and safely accessible cutaneous, subcutaneous, or nodal melanoma lesion >= 5 mm in longest diameter for metastatic cutaneous or mucosal melanoma
  * At least one safely accessible liver metastasis for patients with metastatic ocular melanoma
* Patients with metastatic ocular melanoma must meet all of the additional inclusion criteria:

  * No more than 25% overall tumor involvement of the liver by magnetic resonance imaging (MRI) imaging
  * Child Pugh Score A
  * Absence of ascites
  * No portal vein thrombosis
* Have resolution of all previous treatment-related toxicities to grade 1 severity or lower
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 14 days prior to registration)
* Hemoglobin >= 9.0 g/dL (without need for hematopoietic growth factor or transfusion support) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Aspartate transaminase (AST) =< 2.5 x ULN (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x ULN (obtained =< 14 days prior to registration)
* Prothrombin time (PT) =< 1.5 x ULN (or international normalization ratio [INR] =< 1.4) or partial thromboplastin time (PTT)/activated partial thromboplastin time (aPTT) =< ULN (obtained =< 14 days prior to registration)
* Serum creatinine within institutional limits of normal (=< ULN) (obtained =< 14 days prior to registration)
* Life expectancy of >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Willing and have the ability to comply with scheduled visits (including geographical proximity), treatment plans, laboratory tests, and other study procedures
* Willing to provide all biological specimens as required by the protocol including fresh tissue for biomarker analysis (metastatic melanoma cohort with accessible injectable lesions only)

  * NOTE: Patients with cutaneous melanoma and accessible cutaneous/subcutaneous lesions will have one lesion biopsied prior to the subject receiving the first dose of study treatment on day 1 of cycle 1 and the biopsy will be repeated on the injected target lesion and an uninjected lesion where possible post-virus treatment on day 3
  * NOTE: Repeat samples may be required if adequate tissue is not obtained
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

  * NOTE: if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Willing to use an adequate method of contraception from the first dose of study medication through 120 days after the last dose of study medication, for persons of childbearing potential or persons able to father a child only

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Any of the following prior therapies:

  * Prior chemotherapy =< 2 weeks prior to registration
  * Prior immunotherapy (monoclonal antibodies) =< 3 weeks prior to registration
  * Prior experimental agent =< 2 weeks prior to registration
  * Prior radiation therapy =< 2 weeks prior to registration
* Need for concurrent chemotherapy, immunotherapy, radiotherapy, ablation therapy or any ancillary therapy considered investigational (used for a non-FDA approved indication or in the context of a research investigation)
* Minor surgical or interventional procedure =< 7 days prior to registration
* Major surgical procedure =< 21 days prior to registration
* History or evidence of melanoma associated with immunodeficiency states (e.g., hereditary immune deficiency, organ transplant, or leukemia, requires concomitant treatment with immunosuppressive agents, including CTLA-4 agonists, or chronic oral or systemic steroid medication including physiological replacement doses for adrenal insufficiency
* History of or plan for splenectomy or splenic irradiation
* History or evidence of central nervous system (CNS) metastases
* Active skin lesions (open wounds, severe rash, herpetic lesions, etc.)
* Prior non-oncology vaccine therapies used for the prevention of infectious disease =< 28 days prior to registration
* Requires concomitant treatment with therapeutic anticoagulants
* Known history of active tuberculosis
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Known acute or chronic hepatitis B or hepatitis C infection (requires negative test)
* Metastatic ocular melanoma patients only: liver radioembolization =< 90 days prior to registration
* No other active second malignancy other than non-melanoma skin cancers and in situ cervical cancers within 3 years of registration

  * NOTE: A second malignancy is not considered active if all treatment for that malignancy is completed and the patient has been disease-free for at least 3 years prior to registration
* No uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled symptomatic cardiac arrhythmia
  * Uncontrolled hypertension (defined as blood pressure > 160/90)
* New York Heart Association classification III or IV, known symptomatic coronary artery disease or symptoms of coronary artery disease on systems review, or known cardiac arrhythmias
* Active CNS disorder or seizure disorder or known CNS disease or neurologic symptomatology
* Pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of study treatment
* Person of childbearing potential who is unwilling to use two (2) highly effective methods of contraception during study treatment and through 120 days after the last dose of study treatment
* Person able to father a child who is unwilling to use a highly effective method of contraception during study treatment and through 120 days after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2025-10-12 (Actual); Study Completion 2025-10-12 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose | Up to 28 days
  The maximum tolerated dose is defined as the highest dose level among those tested where at most 1 out of 6 patients develops a dose-limiting toxicity (DLT) prior to the start of their second cycle of treatment and the next highest dose level is such that 2 of the 3 to 6 patients treated at this dose level develop a DLT prior to the start of their second cycle of treatment.
Incidence of adverse events | Up to 42 days after treatment for Group A and 28 days after treatment for Group B
  Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed by dose level to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

SECONDARY OUTCOMES:
Tumor response rate | Up to 1 year
  A tumor response is defined as either a complete response or partial response on two consecutive evaluations at least 6 weeks apart. Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by dose level).
Overall survival | From registration to death due to any cause, assessed up to 1 year
  The distribution of survival time will be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Roxana S. Dronca, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

DOCUMENTS (1):
  • Informed Consent Form (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03865212/ICF_000.pdf